CLINICAL TRIAL: NCT06929312
Title: Effectiveness Of Simulation Based Training Versus Traditional Lecturing For Outbreak Investigation Among Medical Students: A Randomised Control Trial
Brief Title: Simulation Based Training In Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1011/ERC/CMH/LMC; NCT07115264 (obsolete NCT alias)
Record Dates: First submitted 2025-03-17; First posted 2025-04-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cholera
Keywords: Cholera Outbreak Investigation; Cholera; Medical students
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tabletop Simulation Based Teaching (Experimental): A pre tested and validated questionnaire was use tabletop simulation method on cholera outbreak
  Interventions: Other: Tabletop simulation based teaching
- Conventional Class room teaching (Active Comparator): conventional class room lecture was used on cholera outbreak.
  Interventions: Other: conventional class room teaching

INTERVENTIONS:
Other: Tabletop simulation based teaching — a pre tested and validated questionnaire was used as a tabletop simulation method on Cholera outbreak.
  Arms: Tabletop Simulation Based Teaching
Other: conventional class room teaching — conventional class room lecture using power point was delivered on Cholera outbreak.
  Arms: Conventional Class room teaching

SUMMARY:
Transferring classroom learning to real-life situations is a challenge. Tabletop simulation exercises offer a low-cost and context-specific approach for educating students on appropriate responses during health emergencies.

This randomized controlled trial will evaluate the effectiveness of simulation-based training versus traditional lecture methods in enhancing outbreak investigation skills among medical students.

DETAILED DESCRIPTION:
This randomized controlled trial will assess the efficacy of simulation-based training compared to conventional lecture methods in improving medical students' outbreak investigation skills. it will be Conducted at CMH Lahore Medical College over nine months, the trial will include 4th year MBBS students with no prior outbreak investigation training. Participants will be randomized into two groups: an intervention group undergoing simulation-based exercises and a control group receiving traditional lectures.

ELIGIBILITY:
Inclusion Criteria:

* 4th year MBBS students at CMH Lahore Medical College without prior outbreak investigation training,
* willing to participate and providing informed consent.

Exclusion Criteria:

* students with supplementary exams
* unwillingness to participate, or
* scheduling constraints.

Ages: 22 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Outcome will be measured via knowledge, expertise in outbreak investigation, and attitude toward community medicine. | at baseline and after two week of teaching methodology applied
  The primary outcome will be measured using the Cholera Outbreak Investigation Training Questionnaire (COIT-Q)-a self-designed, pre-validated tool that will evaluate:
  Knowledge Domain: 10 MCQs (1 mark each; total = 10 marks)
  Skills Domain: 6 scenario-based items rated 0-2 each (total = 12 marks)
  Attitude Domain: 5 Likert-scale items (1-5 per item; total = 25 marks)

CONTACTS AND LOCATIONS:
Overall Officials: Tahira Raza, Principal Investigator — Department of Community Medicine, CMH Lahore Medical College & IOD (NUMS Rawalpindi)
Locations (1):
- CMH Lahore Medical College and Institute of Dentistry, Lahore, Pakistan